CLINICAL TRIAL: NCT02914834
Title: Feasibility Testing of a Randomized Controlled Trial of Acupuncture to Improve Symptoms for Individuals With Stable Angina (AIMS-A)
Brief Title: Acupuncture for Individuals With Stable Angina
Acronym: AIMS-A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research activity halted due to the Coronavirus Disease 2019 (COVID-19) pandemic. We were obliged to stop the in-person study in March 2020 due to the mandated lockdowns as a result of COVID.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Judith Schlaeger, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0642; R21NR017705-01A1 (NIH)
Record Dates: First submitted 2016-08-13; First posted 2016-09-26 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Angina, Stable; Chest Pain; Microvascular Angina; Heart Failure
MeSH Terms: conditions — Angina, Stable; Chest Pain; Microvascular Angina; Heart Failure | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Acupuncture (Experimental): Standardized acupuncture protocol twice per week for 5 weeks for a total of 10 sessions
  Interventions: Other: Acupuncture
- Non-pain related video health education (Active Comparator): The attention control group will receive non-pain related video health education over 5 weeks equal to the approximate 10 hours of treatment for the acupuncture group.
  Interventions: Other: Non-pain related video health education

INTERVENTIONS:
Other: Acupuncture — Standardized acupuncture treatment administered for 30 minutes each session
  Arms: Device Acupuncture
Other: Non-pain related video health education — Attention control group will watch health education videos the equivalent of 10 hours from randomization up to study completion.
  Arms: Non-pain related video health education

SUMMARY:
This RCT aims to determine if it is possible to perform acupuncture on men and women diagnosed with stable angina who have symptoms, chest pain, and/or chest discomfort. The investigators want to determine if acupuncture reduces the pain and other symptoms of angina, chest pain, and chest discomfort. The investigators also want to examine whether this study is acceptable to the participants, and by carrying out this study the investigators will be able to tell how many participants they will need in a future larger study to further test acupuncture to reduce the symptoms of angina in women.

DETAILED DESCRIPTION:
The investigators are conducting a RCT aimed at gathering feasibility, and initial efficacy for a randomized controlled trial (RCT) to test the effect of acupuncture on anginal symptoms, chest pain, and chest discomfort in men and women. The investigators long term goal is pain and symptom management resulting in improved functional status and quality of life for men and women with stable angina, chest pain, and chest discomfort. This study will include 69 community dwelling men and women with a medically confirmed diagnosis of stable angina, chest pain which includes non-ischemic or ischemic cardiomyopathy, microvascular coronary dysfunction (MCD), heart failure with preserved ejection fraction (HFpEF), heart failure with reduced ejection fraction (HFrEF), or chest discomfort whose pain and associated symptoms have not been completely controlled with guideline-directed medical management. The investigators will use a randomized attention control design with 13 men and women assigned to initial acupuncture and 13 to control. Participants in the experimental group will receive a standardized acupuncture point prescription two treatments per week, for 5 weeks. The attention control group will receive non-pain related video health education over 5 weeks equal to the approximate 10 hours of treatment for the acupuncture group.

ELIGIBILITY:
Inclusion criteria:

* provision of a verified diagnosis from a care provider
* male or female sex
* at least 21 years of age
* intermittent angina symptoms (pain, pressure, or discomfort in the chest or other areas of the upper body)
* medical confirmation of a diagnosis of stable angina for at least 6 months

medical confirmation of a diagnosis of chest pain including non-ischemic or ischemic cardiomyopathy

medical confirmation of a diagnosis of microvascular coronary dysfunction (MCD)

medical confirmation of a diagnosis of heart failure with preserved ejection fraction (HFpEF), heart failure with reduced ejection fraction (HFrEF) medical confirmation of chest discomfort.

Exclusion criteria:

* pregnancy
* chronic obstructive pulmonary disease (COPD) causing pain or associated symptoms
* autoimmune dysfunction
* use of steroid medications
* concomitant physical therapy
* biofeedback
* massage
* additional acupuncture

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holli A DeVon, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeVon HA, Uwizeye G, Cai HY, Shroff AR, Briller JE, Ardati A, Hoppensteadt D, Rountree L, Schlaeger JM. Feasibility and preliminary efficacy of acupuncture for angina in an underserved diverse population. Acupunct Med. 2022 Apr;40(2):152-159. doi: 10.1177/09645284211055754. Epub 2021 Dec 2. PMID 34856826

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Started | 12 | 15
Completed | 11 | 13
Not Completed | 1 | 2
Not completed — Study halted due to COVID | 1 | 1
Not completed — 1 subject withdrew | 0 | 1

BASELINE CHARACTERISTICS:
Population: 27 subjects recruited and enrolled, 24 subjects completed the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 4 | 3 | 7
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Protocol
Description: Feasibility was measured by recruitment (%), retention (%), completion (%). Feasibility was defined as ≥ 80% recruitment, ≥75% retention following enrollment, and ≥ 80% completion.
Time Frame: After 10th acupuncture treatment, at 5 weeks post-baseline (study completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 12 | 15
Participants
  Participants recruited | 12 | 15
  Participants retained | 12 | 15
  Participants completed | 11 | 13

2. Primary Outcome: Protocol Acceptability Scale for Treating Angina With Acupuncture
Description: Protocol Acceptability Scale for Treating Angina with Acupuncture is a 9-item instrument used to measure acceptability of the study processes and protocols. Items are measured on a 0 to 2 scale, where 0 means "did not like the study and did not like acupuncture", and 2 means "liked the study and liked acupuncture". The protocol was deemed to have high acceptability if 80% of participants scored ≥ 80% of possible points on the acceptability scale. The investigators calculated the mean score for each of the 9 questions in each arm, divided the total score for the 9 questions by the maximum possible points for the measure (18 x number of participants in each arm), and converted the total mean scores to percentage of participants who liked the study/liked acupuncture in each arm.
Time Frame: After 10th acupuncture treatment, at 5 weeks post-baseline (study completion)
Population: Those completing the study protocol at 5 weeks
Measure: Number; unit: percentage of subjects who liked study
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 11 | 13
percentage of subjects who liked study | 87.9 | 51.7

3. Secondary Outcome: Average Pain Intensity From the McGill Pain Questionnaire
Description: Average Pain Intensity from the McGill Pain Questionnaire is the average of pain now, least pain in the past 24 hours, and worst pain in the past 24 hours. Average Pain Intensity is scored on a 0 to 10 Likert type scale with 0 = no pain and 10 = excruciating pain. Pain intensity is the pre-specified outcome measure, while pain now and least and worst pain are values used to calculate average pain intensity and were not specified outcome measures.
Time Frame: From before first treatment at baseline to after 10th acupuncture treatment (study completion) at 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 11 | 13
score on a scale
  Baseline Average pain intensity | 3.81 (1.99) | 3.42 (2.56)
  Completion Average pain intensity | 1.21 (1.13) | 2.97 (1.96)

4. Secondary Outcome: Seattle Angina Questionnaire-7 (SAQ-7)
Description: The instrument consists of 7 items measuring functional status, symptoms, and quality of life on participants. Item responses are coded sequentially from worst to best status and range from 1 to 6, except Quality of Life (range 1-5). Scores are generated for each domain and are scaled 0 to 100, with 0 denoting the worst and 100 the best possible status.
Time Frame: From before first treatment at baseline to after 10th acupuncture treatment (study completion) at 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 11 | 13
score on a scale
  Baseline Functional status | 16.67 (15.18) | 29.78 (26.77)
  Completion Functional status | 46.67 (27.49) | 16.92 (19.36)
  Baseline symptoms | 55.00 (20.23) | 62.67 (13.35)
  Completion Symptoms | 72.73 (15.55) | 56.15 (8.70)
  Baseline Quality of Life | 20.83 (26.82) | 16.67 (13.91)
  Completion Quality of life | 54.55 (23.90) | 11.54 (12.97)
  Baseline Total score | 29.29 (13.01) | 36.57 (16.14)
  Completion Total score | 56.44 (19.74) | 27.51 (9.21)

5. Other Pre Specified Outcome: Inflammatory Biomarkers Blood Test
Description: Inflammatory biomarkers between the acupuncture and control group [interleukin (IL)- 2, IL-4, IL-6, IL-8, IL-10, IL-18; tumor necrosis factor alpha (TNF-α)]. Changes in these values from before first treatment at baseline to after 10th acupuncture treatment at 5 weeks is reported.
Time Frame: From before first treatment at baseline to after 10th acupuncture treatment (study completion) at 5 weeks
Population: Overall number of participants analyzed differ based on difficulty drawing blood on subjects.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 6 | 11
pg/ml
  Mean change IL-2 | 0.394 (22.523) | 11.595 (17.414)
  Mean Change IL-4 | -1.444 (2.724) | -.818 (2.306)
  Mean Change IL-6: number analyzed (Participants) | 6 | 10
  Mean Change IL-6 | -.096 (.863) | -.212 (1.224)
  Mean Change IL-8 | 2.065 (7.671) | 1.255 (5.373)
  Mean Change IL-10 | 4.317 (14.373) | 7.386 (38.165)
  Mean Change IL-18 | 55.695 (65.646) | 16.540 (68.665)
  Mean change TNF-alpha: number analyzed (Participants) | 6 | 10
  Mean change TNF-alpha | 6.312 (25.370) | 8.763 (20.667)

6. Other Pre Specified Outcome: Inflammatory Biomarkers Blood Test- Mean Change C-reactive Protein (CRP)
Description: Inflammatory biomarker CRP between the acupuncture and control group. Changes in these values from before first treatment at baseline to after 10th acupuncture treatment at 5 weeks is reported.
Time Frame: From before first treatment at baseline to after 10th acupuncture treatment (study completion) at 5 weeks.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
Number analyzed (Participants) | 6 | 11
ng/ml | -302.903 (1049.445) | -457.205 (1416.052)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over the duration of the 5-week study protocol
Arm/Group | Device Acupuncture | Non-pain Related Video Health Education
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02914834/Prot_SAP_000.pdf